CLINICAL TRIAL: NCT03619967
Title: Sentinel Lymph Node Mapping With Near Infrared Fluorescent Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Ss. Cyril and Methodius University of Skopje, Macedonia (Unknown)
Responsible Party: Principal Investigator, Viktor Gruev, PhD, Professor, University of Illinois at Urbana-Champaign
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18947
Record Dates: First submitted 2018-07-17; First posted 2018-08-08 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; sentynel lymph node; fluorescence imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Experimental: Arm 1: Multispectral Imaging Per current standard of care for patients with breast cancer, three different tracers will be injected in the patient: technetium radiocolloid, indocyanine green and methylene blue. The surgeon will identify the location of the sentinel lymph node per standard of care by using a handheld gamma-probe and by visual inspection of the wound site. During this same time period, fluorescent signals from the underarm surgical wound site will be recorded with the bio-inspired multispectral camera.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multispectral imaging device (Experimental): Bio-inspired multispectral imaging device will be used to record fluorescence signals emited by dyes (Indocyanine green and methylene blue) routinely used for visual identification of sentinel lymph nodes per current standard of care worldwide.
  Interventions: Device: Multispectral imager

INTERVENTIONS:
Device: Multispectral imager — Device: Bio-inspired multispectral imager
  -Manufactured at University of Illinois at Urbana Champaign

SUMMARY:
Surgery is the primary curative option for patients with cancer, with the overall objective of complete resection of all cancerous tissue while avoiding damage to healthy tissue. In addition, sentinel lymph node (SLN) mapping and resection is an essential step in staging and managing the disease. Even with the latest advancements in imaging technology, incomplete tumor resection in patients with breast cancer is at an alarming rate of 20-25%, with recurrence rates of up to 27%. The clinical need for imaging instruments that provide real-time feedback in the operating room is unmet, largely due to the use of imaging systems based on contemporary technological advances in the semiconductor and optical fields, which have bulky and costly designs with suboptimal sensitivity and co-registration accuracy between multimodal images.

To address these challenges, the investigators have introduced an innovative design comprising a bio-inspired multispectral sensor which can significantly improve image-guided surgery. The objective of this clinical study is to determine the feasibility of using a bio-inspired multispectral imaging system to detect sentinel lymph nodes and cancerous tissue during intraoperative procedures in patients with breast cancer.

DETAILED DESCRIPTION:
Per current standard of care for patients with breast cancer, three different tracers will be injected in the participants: technetium radiocolloid, indocyanine green and methylene blue. Initially, the surgeon will identify the location of the sentinel lymph node per standard of care by using a handheld gamma-probe and by visual inspection of the wound site. While the surgeon is locating the sentinel lymph nodes in the underarm surgical wound site, the investigators will be recording the fluorescent signals from the same site with the bio-inspired multispectral camera.

All resected tissue from the patient will be imaged with the multispectral camera before sending samples for pathology analysis. Results obtained from the multispectral cameras will not be presented to the surgeon during the surgery in order not to influence their surgical decision.

ELIGIBILITY:
Inclusion Criteria:

* early or progressive stage of breast cancer
* able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* inflammatory cancerous tissue
* pregnant women
* history of allergic reactions to iodide or seafood allergy
* sentinel lymph nodes were not detected with radiocolloid and static gamma camera
* patients have previous breast surgery
* patients who were unwilling to enter the study

Ages: 17 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Fluorescence imaging of sentinel lymph nodes with indocyanine green and methylene blue. | Up to 1 week after surgery
  The patient will be admitted to the hospital one day before the surgery and will be treated without deviating from normal operating procedures for this surgical procedure. The patient will be first administered radiocolloid tracer per current standard of care and scanned with a double-headed SPECT gamma camera to locate sentinel lymph nodes (SLN).
  The patient is moved to the operating room next. After the patient undergoes anesthesia, methylene blue and indocyanine green will be administered. The surgeon will look to locate radioactive activity and coloration from methylene blue and indocyanine green.
  While the surgeon is locating the SLN in the underarm surgical wound site, the investigators will be recording the fluorescent signals from the same site with the multispectral camera. After the location of the sentinel lymph node, the surgeon will resect this tissue and with a handheld gamma probe will test for accumulation of the radio tracer.

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Gruev, PhD, Principal Investigator — UIUC
Locations (1):
- University Clinic Hospital, Skopje, North Macedonia

IPD SHARING:
Plan to Share IPD: No